CLINICAL TRIAL: NCT02436161
Title: Effectiveness of a Multidisciplinary Care Management Program for High-risk Patients Who Are Admitted at Hospital Because of Heart Failure (PROMIC)
Brief Title: Effectiveness of a Multidisciplinary Care Management Program for High-risk Patients With Heart Failure (PROMIC)
Acronym: PROMIC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Basque Health Service (Other Government)
Responsible Party: Principal Investigator, Cristina Domingo, Family physician, Basque Health Service
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: BG2010111182
Record Dates: First submitted 2015-04-26; First posted 2015-05-06 (Estimated); Last update posted 2015-05-06 (Estimated); Status verified 2015-05

CONDITIONS: Heart Failure
Keywords: Heart Failure; Comorbidity; Patient Care Management; Primary Health Care; Delivery of Health Care, Integrated
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Care management program "PROMIC" (Experimental): care management program provided by a multidisciplinary team that optimizes care with the main role of nurses acting as coaches of patients and carers, within the primary care teams
  Interventions: Behavioral: Care management program "PROMIC"
- Usual care (No Intervention): Patients in the control group belongs to different Primary health care centres from the intervention group and are treated as usual by their Primary Care team and by cardiologists different from the intervention group

INTERVENTIONS:
Behavioral: Care management program "PROMIC" — intensive coaching intervention to optimize care and prevent readmissions, using educational selfcare and worsening symptoms recognition by patients and carers
  Arms: Care management program "PROMIC"

SUMMARY:
OBJECTIVE: To evaluate the effectiveness of a multidisciplinary care management collaborative program for high-risk patients with heart failure (HF) who are admitted at hospital, based on the 6 components of the Chronic Care Model "PROMIC", in terms of reduction of a Combined event rate (readmissions / cardiac events / death / emergency department visits) and other variables, the feasibility of the program, the improvement on quality of life related to health and functional capacity of the PROMIC patients compared with control patients in usual care.

DESIGN: A quasi-experimental, prospective one year follow-up study. SETTING AND SUBJECTS: Primary Health care Centres of Interior County in Bizkaia and of Araba County in Araba, Galdakao Hospital, Santa Marina Hospital and University hospital os Araba in the Basque Country. Will be captured as a minimum intervention group of 125 patients admitted for HF in New York Heart Association (NYHA) functional status II-III-IV from previous mentioned hospitals. Another 125 patients from different primary health care centers, will be the control group.

INTERVENTION: The intervention to be applied will be PROMIC, control patients will receive usual care MEASUREMENTS: The mean outcome measure will be the time free of events from the time of inclusion to the first event (readmission / cardiac events / death / emergency visits). Secondary endpoints will be the quality of life related to health (MLFHQ and SF-12), functional capacity (6-Minute Walk Test), structural changes in cardiac structure (natriuretic peptide levels), adherence to drug treatment (Morinsky-Green), the cost of the program, the usefulness and acceptability of PROMIC by professionals and patients. Predictor variables also will be collected such as sex, age, education level, co-morbidity, social risk level, dependency etc.

STATISTICAL ANALYSIS: Analysis was performed by intention to treat. Survival curves will done. A model of Cox proportional hazards will be built.

DETAILED DESCRIPTION:
INTRODUCTION In light of the increased prevalence of chronic diseases and comorbidities as a result of the increased life expectancy of the population, the need to develop care models that adequately respond to the healthcare and sociodemographic needs of the populatión in the actual context in which they are applied has been proposed. Patients with chronic and/or multiple diseases present the greatest health care needs and tend to experience the imbalances in the system with the greatest intensity. Investigators have concentrated the research on patients admitted because of HF due to the high prevalence and complexity of this disease and the fact that such patients present multiple chronic conditions. These patients are normally elderly and present high degrees of comorbidity and poly-medication, poor treatment adherence and difficulties in selfcare. The majority of patients admitted with HF are in level 3 of the Kaiser pyramid together with other patients with complex health care needs.

There is some evidence that a higher degree of multidisciplinarity results in better team coordinatión and training and more effective care for complex high-risk patients, of which HF patients are a good example.

PROMIC is an organisational care management innovation that provides a comprehensive and integrated approach to patients with a high degree of complexity, in this case, patients admitted with HF.

It promotes the integratión of care in different healthcare settings with the change of the nurses role and self-care training in patients. As such, PROMIC helps to ensure the continuity of patients care in their own environment.

The aim of the innovative care model that PROMIC is intended to provide in high-risk HF patients is to improve health outcomes and to modify the current care model for chronic diseases, thereby serving as the foundation for future interventions targetting other chronic patients with multiple comorbidities and complex health care needs. Indeed, precisely due to the presence of comorbidities in this type of patient, investigators consider coordination with consultants from other specialities to be essential. As HF patients present marked comorbidity, investigators expect that the experience acquired during this project will help them to design interventions that can be broadened to cover all complex chronic patients likely to benefit from a care management programs.

OBJECTIVES

* To evaluate the effectiveness of a multidisciplinary care management collaborative program for high-risk patients with HF who are admitted at hospital, based on the 6 components of the Chronic Care Model "PROMIC", in terms of reduced Combined event rate (readmissions / cardiac events / death / emergency department visits) and other variables, the feasibility of the program, the improvement on quality of life related to health and functional capacity of the PROMIC patients compared with control patients in usual care.
* To understand the opinion of the professionals involved in the process using discussion and consensus methods in order to design the most effective and comprehensive clinical and organisational intervention.

The goal of this project is to establish a sustainable care model for patients admitted with HF that improves their health outcomes. The understanding gained during implementation of this model will lead to further research involving the care of other types of complex chronic patients.

METHODOLOGY DESIGN: A quasi-experimental, prospective one year follow-up study. SETTING AND SUBJECTS: Primary Health care Centres of Interior County in Bizkaia and of Araba County in Araba, Galdakao Hospital, Santa Marina Hospital and University hospital os Araba in the Basque Country. Will be captured as a minimum intervention group of 125 patients admitted for HF in NYHA functional status II-III-IV from previous mentioned hospitals. Another 125 patients from different primary health care centers will be the control group.

INTERVENTION: The intervention to be applied will be PROMIC, control patients will receive usual care.

PROMIC is an organizational innovation comprising a complex intervention containing components supported by scientific evidence from both a content based on clinical practice guidelines, (CPGs) as well as regarding its implementation, which is based on the Chronic Care Model (CCM), developed by Ed Wagner at the McColl Institute (Seattle, USA) in the 1990s. As this is a complex intervention, investigators have selected the theoretical and methodological framework for the design and evaluation of complex interventions in a clinical setting developed by the healthcare and public health services working group of the United Kingdom Medical Research Council (MRC), which comprises four phases.

In phase 0 investigators have undertaken a strategic needs research and evaluation process and a comprehensive literature search regarding the management of HF patients and complex chronic comorbid patients in order to identify and select areas for optimization. Phase 1 comprised the design of the intervention program in collaboratión with professionals from the fields of primary care, hospital and social care, as well as primary researchers and managers, and the piloting of the intervention with a small number of patients and taking into account the actual context in the Basque country public health system where Primary care is very well developed and effective and with a high quality hospital care. The piloting of the intervention was deployed in 15 polymedicated (mean of 11 drugs) patients admitted with HF and multiple comorbidities (mean of six chronic diseases) to confirm its feasibility. This pilot study concluded with positive results and led to the implementation of a quasi-experimental phase 2 trial.

Intervention (PROMIC) was performed in the framework of each of the six components of the CCM.

1. Healthcare organisation. Investigators held 18 joint working sessions involving all components of the multidisciplinary team to establish the content of the clinical care and organisational interventions.
2. Delivery system design. A care management model describing the circuits and communications between healthcare and non-healthcare professionals was defined in these joint sessions.
3. Use of clinical information systems. Investigators use an electronic case history shared by all professionals involved in patient care, which acts as a care record and action reminder.
4. Decision-making support. Investigators have standardised the information contained in the discharge planning report and the communications between professionals in the return home and protocolized the pharmacological treatments indicated in the guidelines. The individual problems presented by each patient are managed with a comprehensive and personalized intervention.

   Investigators have designed a theoretical/practical training plan for all study participants 27 hours for physicians and 42 hours for nurses, which has been complemented with a course on electrocardiography, basic recommendations for cardiology and drug titration for nursing staff.
5. Education about self-care and empowerment of patients and their families. Creation of a new nursing role aimed at coaching and educating patients and their families and evaluating their level of understanding and self-care. Investigators have prepared educational support material for personalized self-care aimed at patients and their carers.
6. Integration of community resources. Investigators have established meetings and contacts with social workers and community pharmacists.

MEASUREMENTS: The mean outcome measure will be the time free of events from the time of inclusion to the first event (readmission / cardiac events / death / emergency visits). Secondary endpoints will be the quality of life related to health (MLFHQ and SF-12), functional capacity (6-Minute Walk Test), structural changes in cardiac structure (brain natriuretic peptide BNP), adherence to drug treatment (Morinsky- Green questionaire), the cost of the program based in the adjusted clinical group (ACG) , the usefulness and acceptability of PROMIC by professionals and patients. Predictor variables also will be collected such as sex, age, education level, co-morbidity, social risk level and dependency

baseline 6ºmonth 12º month

MLFHQ X X X

SF-12 X X X

6-Minute Walk Test X X X

BNP levels X X X

Morinsky-Green X X X

HFSBS X X X

Charlson Index X X X

Memory impairment Screen (MIS)X X X

HAD (<70years) X X X

Yesavage(>70years) X X X

Duke X X X

Lawton y Brody X X X

Barthel X X X

Zarit X X X

Social evaluation scale X X X

Professional focus group X

Cost X

Perception of integrated care D'Amour X

STATISTICAL ANALYSIS: Analysis was performed by intention to treat. Survival curves will done. A model of Cox proportional hazards will be built.

ELIGIBILITY:
Inclusion Criteria:

* Patients admitted at hospital because of HF in II to IV NYHA stage

Exclusion Criteria:

* life expectancy below 3 months
* discharge to nursing home
* Severe cognitive impairment

Min Age: 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 250 (Actual)
Dates: Start 2011-05; Primary Completion 2013-05 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Hospital readmissions because of HF | one year

SECONDARY OUTCOMES:
Quality of life measured by Minnesota Questionaire and SF12 Questionaire | one year
self management knowledge measured by the Heart Failure Self Behaviour Scale | one year
Cost of the program | one year
professional perception of integrated care measured by the D'Amour Questionaire | one year

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Domingo, MD, FAM PHY, Principal Investigator — Basque Health Service

REFERENCES:
- See also: phase 0 and 1 of the PROMIC care management program — http://www.osakidetza.euskadi.net/contenidos/informacion/2014_osteba_publicacion/es_def/adjuntos/pro_Insufcardio.pdf